CLINICAL TRIAL: NCT02201290
Title: An Extension Study of Eltrombopag in Pediatric Patients With Chronic Immune (Idiopathic) Thrombocytopenia Purpura (ITP)
Brief Title: A Long-term Safety Study of Eltrombopag in Pediatric Patients With Chronic Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 117366; CETB115BRU01 (Other: Novartis); 2017-004082-27 (EudraCT Number)
Record Dates: First submitted 2013-06-06; First posted 2014-07-28 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: Chronic immune thrombocytopenic purpura, ITP, eltrombopag olamine, thrombopoietin receptor agonist, pediatrics
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Intervention Model Description: AEs were graded using the common toxicity criteria for adverse events (CTCAE) Version 4.03. If a patient reported more than one AE with the same preferred term (PT), the AE with the greatest severity was presented. If a patient reported more than one AE within the same primary system organ class (SOC), the patient was counted only once with the greatest severity at the SOC level, where applicable. An AE with missing CTCAE grade was included in the 'All grades' column of the summary tables.
  In AE summaries, the primary SOC was presented alphabetically and the PTs were sorted within the primary SOC in descending frequency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental): Eligible subject will be allocated to 1 of 3 age-defined cohorts. Cohort 1: between 12 and 17 years old, Cohort 2: between 6 and 11 years old, and Cohort 3: between 1 and 5 years old. For Cohorts 1 and 2, eltrombopag tablets will be administered, however, subjects in Cohort 2 may use eltrombopag powder for oral suspension (Eltrombopag PfOS) if they have difficulty swallowing tablets and are receiving a dose of eltrombopag of < 40 mg. For Cohort 3, either eltrombopag tablets or PfOS will be administered.
  Interventions: Drug: Eltrombopag Tablets; Drug: Eltrombopag PfOS

INTERVENTIONS:
Drug: Eltrombopag Tablets — Eltrombopag tablets will be white, round film coated tablets containing eltrombopag olamine equivalent to 12.5 mg, 25 mg, 50 mg and 75 mg of eltrombopag. The 12.5 mg tablet will be smaller than the 25 mg, 50 mg and 75 mg tablets. Subjects will receive maximum dose of 75 mg once daily (QD).
Drug: Eltrombopag PfOS — Eltrombopag PfOS is a reddish-brown to yellow powder contained inside an elongated sachet. Each sachet will contain eltrombopag olamine equivalent to 20 mg of eltrombopag per gram of powder. Subjects will receive maximum dose of 75 mg once daily (QD)

SUMMARY:
This was an open-label Phase III extension study to evaluate the long-term safety of eltrombopag in pediatric patients with chronic ITP who previously participated in study TRA115450. This study allowed dosing of eltrombopag at an individualized dose for each subject based upon platelet count. The starting dose was based on the subject's dose at the end of the TRA115450 study. The maximum dose was 75 mg daily.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from the subject's guardian and accompanying informed assent from the subject (for children over 6 years old).
* Subjects must be between 1 year and <18 years of age at Day 1.
* Subjects must have enrolled in TRA115450/PETIT2 study.
* Subjects must have completed Part 1 and Part 2 of TRA115450/PETIT2 study.
* Female subjects of child-bearing potential (after menarche) must have a negative pregnancy test within 24 hours of first dose of study treatment; agree and be able to provide a blood or urine specimen for pregnancy testing during the study; agree to use effective contraception during the study and for 28 days following the last dose of study treatment, and not be lactating.
* Male subjects with a female partner of childbearing potential must agree to use effective contraception from 2 weeks prior to administration of the first dose of study treatment until 3 months after the last dose of study treatment.

Exclusion Criteria:

* Subjects with any clinically relevant abnormality, other than ITP, identified on the screening examination or any other medical condition or circumstance, which in the opinion of the investigator makes the subject unsuitable for participation in the study or suggests another primary diagnosis (e.g. Thrombocytopenia is secondary to another disease).
* Any subject considered to be a child in care, defined as one who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. This can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a child in care does not include a child who is adopted or who has an appointed legal guardian.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Russia (3):
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 patients received Eltrombapag treatment during the extension study. Four patients (44.4%) completed the study while 5 patients (55.6%) discontinued from treatment and withdrew from the study.
Groups:
- Eltrombopag: treated participants
Period: Overall Study
Arm/Group | Eltrombopag
Started | 9
Completed | 4
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Eltrombopag: all treated participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (3.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Frequency of all adverse events (including Ophthalmic events) categorized using CTCAE toxicity grades and clinical laboratory test [ Time Frame: Up to Week 4 Follow-up period ] Clinical laboratory assessments and frequency of all adverse events, categorized using Common Terminology Criteria for Adverse Events (CTCAE) toxicity grades will present safety and tolerability endpoints
  Serious Adverse Events are below. See All Adverse Events in the following section for specifics
  No statistical analysis was planned for this primary outcome
Time Frame: Up to week 4 follow up period
Population: All treated subjects
Measure: Number; unit: participants
Groups:
- Eltrombopag: Adverse events by system organ class and maximum severity for all treated participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 9
participants
  Number of subjects with at least one event | 3
  Scleral haemorrhage | 1
  Autoimmune hepatitis | 1
  Epistaxis | 1

ADVERSE EVENTS:
Time Frame: up to week 4
Groups:
- Eltrombopag: Eltrombopag was provided to sites by GlaxoSmithKline as tablets or as dry powder for oral suspension (PfOS) sachets
Arm/Group | Eltrombopag
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=9)
Scleral haemorrhage (Eye disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=9)
Nasopharyngitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT02201290/SAP_000.pdf
  • Study Protocol (2013-07-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT02201290/Prot_001.pdf